CLINICAL TRIAL: NCT01348269
Title: A Prospective, Bi-centric,Randomized, Primary Double-blind, Placebo-controlled Phase III Study to Assess the Efficacy of Zoledronic Acid in the Treatment of Bone Marrow Edema Syndrome
Brief Title: Assessment of Efficacy of Zoledronic Acid in the Treatment of Bone Marrow Edema Syndrome
Acronym: ZoMARS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: Crolll Gmbh (Other); University of Wuerzburg (Other)
Responsible Party: Principal Investigator, Dr. Lothar Seefried, Dr. Lothar Seefried, Orthopaedische Klinik Koenig-Ludwig-Haus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446HDE38T
Record Dates: First submitted 2011-05-02; First posted 2011-05-05 (Estimated); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Bone Marrow Edema
Keywords: bone marrow edema; Aclasta
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aclasta (Active Comparator)
  Interventions: Drug: Aclasta
- NaCl Solution (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclasta — 1 x intravenous non-current drip (infusion)
  Arms: Aclasta
Drug: Placebo — NaCl Solution
  Arms: NaCl Solution

SUMMARY:
The primary aim is to test the reduction of bone marrow edema syndrome after a singular intravenous treatment with Zoledronic Acid within 6 weeks compared to placebo. The volume of the edema is defined as biometric data measured by the use of MRT before and six weeks after treatment. The hypothesis has to be checked whether Zoledronic Acid is efficient in the treatment of painful bone marrow edema. A statistically significant reduction of the edema in the MRT is considered as evidence for efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Men: age over ≥ 18 years or women: age over ≥ 18 years with finished reproductivity according to the following definition:
* ≥ 12 month persistent natural (spontaneous) amenorrhoea (women aged <50: additionally: FSH >40MIE/ml and estrogen deficiency of <30pg/ml or a negative estrogen test)
* status post hysterectomy and / or bilateral oophorectomy
* finished reproduction planning
* secure diagnosis of bone marrow edema using MRT
* current osteologic basic laboratory values (≤ 4 weeks before V2) according to DVO criteria
* presence of an personally signed informed consent for the participation in the study

Exclusion Criteria:

* - subchondral bone loss or already occurred cartilage damage due to the bone marrow edema
* reactive bone marrow edema with advanced arthrotic changes in the adjacent joint (grade III and IV according to Kellgren and Lawrence)
* patients with edematous changes in bone marrow due to the diagnosis of M. Sudeck / algodystrophy / Complex Regional Pain Syndrome (CRPS)
* patients with known hypo- and hyperparathyroidism, osteogenesis imperfecta, osteomalacia, M. Paget or another systemic skeletal diseases, except osteoporosis
* patients with bone necrosis in the painful skeletal region
* patients with infectious process at the affected bone or the adjacent joint and adjacent soft parts, respectively
* patients with diagnosed or assumed rheumatoid arthritis, Lupus erythematodes, collagenosis or vasculitides
* patients with advanced renal insufficiency (GFR according to Cockcroft

  / Gault ≤ 40 ml/min/KO)
* patients with malignant diseases with osseous manifestation in anamnesis/history
* status post malignant basic/primary disease with large dosed chemotherapy
* current or massive dose therapy completed before less than 6 weeks (>7.5mg prednisolon equivalent) with glucocorticoids
* patients with a malignant tumor disease within the past 5 years, independent from the affected organ system and independent from the implemented treatment, the presence of a relapse or metastatic invasion, except basal cell carcinoma and squamous-cell carcinoma of the skin Current treatment due to uveitis
* vague/ambiguous hyper- or hypocalcemia, hyper- or hypophosphatemia
* etiological vague/ambiguous AP-increase
* symptomatic renal calculus or nephrocalcinosis within 2 years before V2
* recent fracture within the last 3 months independent of the localisation
* non consolidated fractures
* previous treatment with i.v. bisphosphonates within the last 12 months
* previous treatment with oral bisphosphonates within the last 12 months and longer than 3 months
* pre-treatment with prostacyclin analogs (Ilomedin® / Iloprost®) within the past 6 months
* Current treatment due to inflammatory diseases of the jaw area as well as planned tooth extractions or tooth extractions less than 6 months ago or oral surgery implant treatment
* pregnancy or nursing period
* patients immediately involved in the conduction of the trial and relatives
* patients with current proceedings related to the bone marrow edema
* patients for which the participation in the study carries an increased risk under consideration of the health condition due to the assessment of the investigator
* participation in another clinical trial within 30 days before study start or during the trial
* participation of patient who might be dependent on the investigator, also the spouse, parents or children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2015-08-26 (Actual); Study Completion 2015-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Meffert, Prof. Dr., Study Chair — Department of trauma, hand, reconstructive and plastic, University of Wuerzburg
Locations (2):
- Germany (2):
  - Orthopedic Center for Musculoskeletal Research, Orthopedic Department, University of Wuerzburg, Würzburg, Bavaria
  - Department of trauma, hand, reconstructive and plastic, University of Wuerzburg, Würzburg, Bavaria

RESULTS

PARTICIPANT FLOW:
Groups:
- Zoledronic Acid: single-dose zoledronic acid (Aclasta) with vitamin D 1000IU/d - 5 mg i.v.
- Placebo: placebo with vitamin D 1000 IU/d (NaCl Solution)
Period: Baseline
Arm/Group | Zoledronic Acid | Placebo
Started | 34 | 14
Completed | 34 | 14
Not Completed | 0 | 0
Period: Treatment | Core Study (Until Week 6)
Arm/Group | Zoledronic Acid | Placebo
Started | 34 | 14
Completed | 34 | 14
Not Completed | 0 | 0
Period: Follow-up (Until Week 12)
Arm/Group | Zoledronic Acid | Placebo
Started | 34 | 14
Completed | 32 | 13
Not Completed | 2 | 1
Not completed — Surgical intervention - not study related | 1 | 0
Not completed — Subsequent follow-up treatment required | 0 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Placebo | Total
Number analyzed (Participants) | 34 | 14 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 13 | 42
  >=65 years | 5 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 22 | 10 | 32
Severity of disease [Count of Participants; unit: Participants]
  mild | 4 | 2 | 6
  moderate | 22 | 10 | 32
  severe | 8 | 2 | 10
Pain (VAS) [Mean (Standard Deviation); unit: units on a scale] — Unidimensonal scale to rate pain. Range 0-100. Higher values indicate more pain.
  units on a scale | 36.9 (27.4) | 34.1 (21.1) | 34.9 (24.8)
Qualeffo-41 [Mean (Standard Deviation); unit: units on a scale] — Quality of life questionnaire in patients with fractures. Answers are standardized so that 1 represents the best and 5 (or 3, or 4) represents the worst quality of life. Lower values indicate better quality of life.
  units on a scale | 2.1 (0.5) | 2.2 (0.6) | 2.1 (0.5)
Subjective estimation of medical condition (Paian Disability Index) [Mean (Standard Deviation); unit: units on a scale] — Pain Disability Index (PDI) is an instrument to measure the impact that pain has on the ability of a person to participate in life activities. Score range 0-70 with higher values indicating greater disability due to pain.
  units on a scale | 20.8 (6.8) | 21.3 (6.4) | 20.8 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: Reduction of the Edema Area
Description: The volume of the edema in cm³ is defined as biometric data measured by the use of MRI before and six weeks after treatment. Edema volume at screening was set to 100%. Edema volume six weeks after study drug administration was provdied as percentage reduction compared to the value at screening
Time Frame: Week 6 after administration of a single intravenous dose of zoledronic acid (5 mg)
Measure: Mean (Standard Deviation); unit: percentage of edema volume
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 13
percentage of edema volume | 64.53 (41.92) | 23.97 (46.52)
Statistical Analysis 1: Comparison: Zoledronic Acid vs Placebo; Test type: Other — T-test (with MITT, omitting outlier value of one patient in placebo group); p = 0.006, t-test, 2 sided
Statistical Analysis 2: Comparison: Zoledronic Acid vs Placebo; Test type: Other — Mann-Whitney-Test; p = 0.015, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Reduction of Pain (VAS)
Description: Reduction of pain as measured by a Visual Analog Scale (VAS). Range 0-100 with higher values indicating worse pain.
Time Frame: Assessment at week 3
Population: Reporting group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
units on a scale | 25.5 (22.7) | 25.6 (24.4)

3. Secondary Outcome: Reduction of Pain
Description: Reduction of pain as measured by a visual analog scale (VAS). Range 0-100. Higher values indicating worse pain.
Time Frame: Assessment at week 6
Population: Reporting group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
units on a scale | 25.0 (28.7) | 38.5 (30.2)

4. Secondary Outcome: Quality of Life (Qualeffo-41 Questionnaire)
Description: Quality of life as measured by the Qualeffo-41 questionnaire - a quality of life questionnaire in patients with fractures of the European Foundation for Osteoporosis Higher values indicate worse quality of life
Time Frame: Assessment at week 3
Population: Reporting group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
units on a scale | 2.1 (0.4) | 2.1 (0.6)

5. Secondary Outcome: Quality of Life (Qualeffo-41 Questionnaire)
Description: Quality of life as measured by the Qualeffo-41 questionnaire - a quality of life questionnaire in patients with vertebral fractures of the European Foundation for Osteoporosis
Time Frame: Assessment at week 6
Population: Reporting group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
units on a scale | 2.0 (0.5) | 2.1 (0.6)

6. Secondary Outcome: Subjective Estimation of Medical Condition (PDI)
Description: Subjective estimation of medical condition as assessed by PDI (Pain Disability Index). Range 0-70. The higher the index the greater the person's disability due to pain.
Time Frame: Assessment at week 3
Population: Reporting group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
units on a scale | 14.8 (5.8) | 20.5 (7.3)

7. Secondary Outcome: Subjective Estimation of Medical Condition (PDI)
Description: Subjective estimation of medical condition as assessed by PDI (Pain Disability Index)
Time Frame: Assessment at week 6
Population: Reporting group
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
units on a scale | 13.1 (6.0) | 18.8 (7.7)

8. Secondary Outcome: Number of Additional Medicinal Visits
Description: Number of additional medicinal visits until week 3
Time Frame: Assessment at week 3
Population: Reporting group
Measure: Number; unit: Number of additional medicinal visits
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
Number of additional medicinal visits | 1 | 0

9. Secondary Outcome: Number of Additional Medicinal Visits
Description: Aggregated number of unscheduled medicinal visits
Time Frame: Assessment at week 6
Population: Reporting Group
Measure: Number; unit: Medicinal Visits
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
Medicinal Visits | 0 | 0

10. Secondary Outcome: Number of Days of Illness
Description: Aggregated number of days of illness i.e. sick leave from work, assessed until week 6
Time Frame: Assessment at week 6
Population: Reporting group
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
days | 1.24 (5.02) | 3.00 (7.63)

11. Secondary Outcome: Number of Days of Illness
Description: Number of days of illness assessed until week 6
Time Frame: Assessment at week 6
Population: Reporting group
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
days | 0.94 (4.10) | 3.14 (4.10)

12. Secondary Outcome: Number of Aseptic Bone Necrosis and Fatigue Fractures
Description: Assessment of number of patients withaseptic bone necrosis and/or fatigue fractures.
Time Frame: Baseline until end of study (week 12)
Population: Reporting group
Measure: Count of Participants; unit: Participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: including changes in the following parameters according to DVO guidelines: Calcium, Phosphate, Creatinin-Clearance (Cockcroft-Gault), Alkaline Phosphatase, γGT, CRP
Time Frame: Week 3, 6
Population: Reporting Group
Measure: Number; unit: participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 14
participants
  Serum Calcium | 0 | 0
  Serum Phosphate | 0 | 0
  Serum Alkaline Phosphatase | 0 | 0
  Gamma-GT | 0 | 0
  Serum Creatinine | 0 | 1
  C-reactives protein | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from time of enrollment until completion of follow up, i.e. for 12 weeks
Arm/Group | Zoledronic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/14
Serious Adverse Events (participants affected / at risk) | 4/34 | 1/14
Other Adverse Events (participants affected / at risk) | 34/34 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=34) | Placebo (N=14)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=34) | Placebo (N=14)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (34) | 0 (0)
Chills (General disorders) | 8 (8) | 2 (2)
Fatigue (General disorders) | 10 (11) | 3 (3)
Influenza like illness (General disorders) | 3 (3) | 2 (3)
Malaise (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 13 (14) | 5 (6)
Sciatica (Nervous system disorders) | 1 (1) | 1 (1)
Blepharospasm (Eye disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Renal pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (11) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (4) | 2 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No